CLINICAL TRIAL: NCT04541056
Title: The Effect of Goal Management Training for Adult Survivors of Childhood Leukemia and Non-Hodgkins Lymphoma With Neurocognitive Sequelae: A Randomized Controlled Trial
Brief Title: Goal Management Training for Adult Survivors of Childhood Leukemia and Non-Hodgkins Lymphoma With Neurocognitive Sequelae
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Oslo University Hospital (Other); Norwegian Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/1810
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Childhood Non-Hodgkin Lymphoma; Childhood Acute Lymphoblastic Leukemia; Childhood Acute Myeloid Leukemia
Keywords: Adult survivor; Childhood; Cognitive Remediation; Executive Function; Cognitive Rehabilitation; Cognitive Training; Metacognitive; Late effects; Goal Management Training; Cancer
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal Management Training (GMT) (Experimental): GMT will be administrated in a group-based format over 5 sessions (minimum three weeks between each session). Homework assignments between sessions are included. Following the fourth session, text messages reading "Stop!" (a key instruction in GMT) will be sent to all GMT participants every day to maximize adherence to training (approximately 12 per participant). Homework assignment will also include the logging of automatic thoughts and an examination of the relationship between situations, thoughts, and accompanying emotions.
  Interventions: Behavioral: Goal Management Training (GMT)
- Waitlist/Brain Health Workshop (BHW) (Active Comparator): The adults participating in the control condition will approximately one year from waitlist, be offered a psycho-educative training program, the BHW, in groups aimed at providing a better understanding of cognitive sequelae after treatment for childhood ALL. BHW will be administrated in a group-based format over 5 sessions (minimum three weeks between each session). Homework assignments between sessions are included. Homework assignments between sessions are included.
  Interventions: Behavioral: Brain Health Workshop (BHW)

INTERVENTIONS:
Behavioral: Goal Management Training (GMT) — The manual comprises an introduction to GMT for the survivors of ALL, and a detailed session structure incorporating cognitive and behavioral tasks. The GMT program involves teaching the participants about goals, attention slips and how to manage these, how to review and prioritize goals (e.g., Stop, Think, Organize, Plan), and how to keep goals in mind (e.g., using analogies such as the mental blackboard). Each session will follow the same general format; namely, facility-delivered presentations, flipchart discussions, group activities and homework.
  Arms: Goal Management Training (GMT)
Behavioral: Brain Health Workshop (BHW) — BHW is a psycho-educative control condition, and is typically part of psycho-educative Acquired Brain Injury (ABI) rehabilitation programs, but adjusted for the ALL group of participants. The psycho-educative control condition BHW will be matched GMT for amount of training and therapist contact. Homework assignment and in-session tasks included readings, brain games, puzzles, and practical exercises such as logging sleep.
  Arms: Waitlist/Brain Health Workshop (BHW)

SUMMARY:
Survivors of childhood cancer are at risk for developing neurocognitive sequelae. Multiple meta-analyses demonstrate significant deficits in overall intellectual abilities, academic functioning and specific cognitive skills among survivors of childhood cancer treated with intrathecal chemotherapy only and/or cranial irradiation. Preventing neurocognitive deficits is therefore of great importance. Unfortunately, intervention studies for this group of survivors are scarce. The main aim of this randomized controlled trial is to determine the efficacy of Goal Management Training (GMT) as a group-based treatment program for 60 adult survivors of childhood leukemia, and non Hodgkins lymphoma, diagnosed between 1980 and 2017 at an age below 18, with attention and executive function deficits. The participants will be randomized to one treatment group (GMT), and one waitlist condition followed by one active control intervention, the "Brain health workshop" (BHW), which has a psycho-educative approach. The follow-up time from diagnosis will be ≥5 years and the age at survey 18-40 years. The study will expand the knowledge base on treatment factors important in improving cognitive function. Results from this study can be implemented in rehabilitation for the young adult survivors of childhood leukemia, and non Hodgkins lymphoma, which will be of importance for their future educational and work-related functioning.

DETAILED DESCRIPTION:
Effect of the GMT/waitlist conditions will be assessed through self-reported and objective measures of neuropsychological function, quality of life and health measurements. To avoid extra training effects of neuropsychological testing on participants allocated to waitlist/BHW, assessment following BHW (approximately one-year post T1) will consist of self-report measures only. Patients in all groups will be reassessed within 14 days post intervention (T2), and at 6 months post intervention (T3).

ELIGIBILITY:
The Norwegian Cancer Registry will identify participants based on the following criteria:

* Acute Lymphoblastic Leukaemia (ALL), Acute Myelogen Leukemia (AML), non Hodgkins Lymphoma diagnosed between 1980 - 2017
* Age when diagnosed <18 år (0-17years)
* Age at survey 18-40 years
* Born between 1980 - 2004
* Minimum five years (≥5) post ALL, AML, NHL diagnosis
* ALL, AML, NHL treatment at Oslo University Hospital and St. Olavs Hospital

Inclusion Criteria

Screening/baseline:

* Written informed consent
* ≥5 years from diagnosis
* Age 18-40
* Without cancer recurrence the last five years
* Understand and speak Norwegian

Additional inclusion criteria for the intervention:

* Experiencing executive dysfunction as determined by a semi-structured interview
* Cognitive capacity to engage with the training, and General Ability Index (GAI) Score ≥70 measured by Wechsler Intelligence Scale for Adults (WAIS-IV)

Exclusion Criteria:

* Cancer recurrence within the last five years
* A history of premorbid Central Nervous System (CNS) injury or disease (e.g., Traumatic brain injury with noticeable cognitive changes, loss of consciousness or injury discovered on CT or MR)
* Pre-existing attention deficit hyperactivity disorder (ADHD)
* Motor or sensory damage impeding study participation
* A major psychiatric disease and/or ongoing substance abuse impeding study participation
* Present suicidal ideation
* Down syndrome

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The Behavior Rating Inventory of Executive Function, Adult (BRIEF-A) | 6 months
  The BRIEF-A self-report questionnaire consists of 75 items on which the patient's symptoms are rated on a 3-point Likert scale. The questionnaire provides a Global Executive Composite (GEC) score (range 75-225) and two index scores: the Behavioral Regulation Index (BRI) (range 30-90) and the Metacognitive Index (MI) (range 40-120). Nine subscales are also provided: Inhibit (range 8-24), Shift (range 6-18), Emotional control (range 10-30), Self-monitor (range 6-18), Initiate (range 8-24), Working memory (range 8-24), Plan/organize (range 10-30), Task monitor (range 6-18) and Organization of materials (range 8-24). Higher scores indicate more executive difficulties. Raw scores are transformed into t scores (M=50, SD=10).

SECONDARY OUTCOMES:
Conner's Continuous Performance Test (CPT-3) | 6 months
  The CPT 3 is a measure of inattention, impulsivity, sustained attention and vigilance. The test is computer based and lasts approximately 14 minutes. The participant is instructed to press the space bar/computer mouse when letters appear, but not when Xs appear on the screen. Higher scores reflect worse performance, and raw scores are converted to T-scores (M=50, SD=10). However, scores will be recoded so that higher scores equal better performance/lower scores equal worse performance.
The Color-Word Interference Test (CWI), from Delis Kaplan Executive Function System | 6 months
  The CWI is a measure of inhibition and cognitive flexibility. The test consists of four conditions; color naming (condition 1), word reading (condition 2), inhibition (condition 3) and inhibition switching (condition 4). Scores are computed for completion time (condition 1-4) and total errors (condition 3 and 4). Higher scores reflect better performance, and raw scores are converted to scaled scores (M=10, SD=3).
The Trail Making Test (TMT): from Delis Kaplan Executive Function System | 6 months
  The TMT from Delis Kaplan Executive Function System is a measure of flexibility/shifting. The primary measure is condition 4 where the participant is asked to shift between number and letter sequencing. The test also measures the basic abilities of visual scanning (condition 1), number- and letter sequencing combined with drawing a line (condition 2 and 3) and motor pace (Condition 5). Scores reflect completion time and raw scores are converted to scaled scores (M=10, SD=3). Higher scores reflect better performance.
California Verbal Learning Test (CVLT II) | 6 months
  The CVLT II a measure of verbal learning and memory. Participants are asked to recall words from list A, both with and without an interruption list B. There are three types of conditions; the participant is asked to freely recall items (free recall), to recall after a cue is presented (cued recall) and to recognize previously presented words (recognition condition). Both short and long delay is measured. Raw scores are converted to Z-scores (M=0, SD=1) and T-scores (M=50, SD=10). Higher scores reflect better performance, except for error measures. For T2 (14 days) follow up, CVLT II Alternative Form will be used.
Wisconsin Card Sorting Test (WCST-64) | 6 months
  The WCST-64 is a measure of abstract thinking and set-shifting/ mental flexibility. The participant is instructed to sort cards according to varying principles. A computer-based version will be employed. Raw scores are converted to T-scores (M=50, SD=10) and higher scores reflect better performance.
The Hotel Task | 6 months
  The Hotel Task is a measure of executive components: planning, organization, self-monitoring and cognitive flexibility. The participant is asked to try out as many as possible of five tasks within a relatively short (15 minutes) time period. Raw scores are computed. Higher scores reflect better performance, except for deviation of optimal time use. The test has been demonstrated to have high ecological validity and ability to detect frontal lobe dysfunction.
The Dysexecutive Questionnaire (DEX - self-report) | 6 months
  The DEX - self-report is a measure of everyday problems with executive function. The questionnaire consists of 20 items with a 5-point Likert scale where the respondent is asked to rate the frequency of cognitive difficulties from 0 (never) to 4 (very often). A higher total score reflects worse executive functioning.
Wechsler Adult Intelligent Scale-IV - Fourth Edition (WAIS-IV) | 6 months
  The subtests: Digit span, letter-number sequencing performance will be used as a measure of Verbal working memory/attention (Working memory index).

OTHER OUTCOMES:
The Pediatric Quality of Life Inventory (PedsQLTM4.0) young adult version | 6 months
  The PedsQLTM4.0 is a measure of health-related quality of life. The 23-item PedsQL, version 4.0 Generic Core Scales, can be grouped into 4 domains of HRQOL: 1) Physical Functioning (8 items), 2) Emotional Functioning (5 items), 3) Social Functioning (5 items), and 4) School Functioning (5 items). In addition to the four subscales, a Total Summary Health score (23 items) can be computed.
The Hopkins Symptom Check List (HSCL-25) | 6 months
  The HSCL-25 is a measure of mental health. The Hopkins Symptom Check List (HSCL-25) is a 25-item self-report measuring adult mental health symptoms within the previous week. Total sum scores range from zero (least symptomatic) to 100 (most symptomatic). A mean item score can also be calculated, in which 1,75 is a common clinical cut-off score. The HSCL-25 is a short version of the HSCL-90.
The General Perceived Self-Efficacy Scale (GPSS) | 6 months
  The GPSS is a measure of self-efficacy. The General Perceived Self-Efficacy Scale (GPSS) is a 10-item psychometric scale assessing the strength of an individual's beliefs in his/her ability to respond to controlled environmental demands and challenges. Items are rated on a 4-point Likert scale (1=not at all true to 4=exactly true). There is no cut-off score on this scale. However, the weighted variance equaled 25.91. Thus, a raw score of 24 is 1 SD below the weighted mean using T-norms from the German version.
The Fatigue Severity Scale (FSS) | 6 months
  The FSS is a measure of fatigue. The Fatigue Severity Scale (FSS) includes nine questions related to how fatigue interferes with certain activities; symptom severity is rated on a 7-point Likert scale (1=strongly disagree to 7=strongly agree). Based on previous reports on the prevalence of fatigue, an FSS score ≥5 is to be interpreted as indicative of severe fatigue.
Fatigue questionnaire (FQ) | 6 months
  The FQ is a measure of fatigue. The FQ is an 11-item questionnaire, assessing physical (items 1-7) and mental (items 8-11) symptoms of fatigue, along with a total score. All items are rated using a 4-point Likert scale (0 = better than usual, 1= no more than usual, 2 = much worse than usual. Fatigue "caseness" is defined by total dichotomized scores >4 and a duration of ≥6 months.
The Resilience Scale for Adults (RSA) | 6 months
  The RSA includes 33 questions related to protective factors. Resilience is rated on a scale from 1 to 7, and a total score reflects degree of resilience. The higher the score on RSA scale, the more protective factors an individual is assumed to have, e.g., better psychological health, and thus, the individual seems to cope better with adverse life events. RSA consists of six factors divided into 1) intrapersonal resources ("Perception of self", "Planned future", "Social competence" and "Structured style"), and 2) interpersonal resources ("Family cohesion" and "Social resources").
Epworth Sleepiness Scale (ESS) | 6 months
  The ESS is a measure of general level of daytime sleepiness. The measure includes 8 items, with scaled scores from 0 (would never doze) to 3 (high chance of dozing), participants are asked to rate their usual chances of dozing off or falling asleep in 8 different situations or activities- The reference range of "normal" ESS scores is zero to 10, while scores of 11-24 represent increasing levels of "excessive daytime sleepiness" (i.e., 0-5: Lower Normal Daytime Sleepiness, 6-10: Higher Normal Daytime Sleepiness, 11-12: Mild Excessive Daytime Sleepiness, 13-15: Moderate Excessive Daytime Sleepiness, 16-24: Severe Excessive Daytime Sleepiness). We will use ESS total score ≥13 as a clinical cut-off.
The Insomnia Severity Index (ISI) | 6 months
  The ISI is a 7-item questionnaire is assessing the nature, severity, and impact of insomnia over the past month. A 5-point Likert scale (0 = none; 4 = very severe) is used to rate each item, with total scores ranging from 0-28 (Total score categories; 0-7; No clinical significant insomnia, 8-14: Subthreshold insomnia, 15-21: Clinical insomnia (moderate severity), 22-28 = Clinical insomnia (severe). We will use the ISI total score ≥15 as a clinical cut-off.
PROMIS Pain Interference (PPI) | 6 months
  The PPI is part of the Patient Reported Outcomes Measurement Information System (PROMIS) and includes 8 items. Pain interference refers to the degree to which pain limits or interferes with the persons physical, mental, and social activities. Items range from 1 "not at all" to 5 "very much". An additional item asks the participant to rate average pain intensity for the last 7 days on another scale ranging from 1 "no pain" to 10 "worst pain imaginable".
Brief Pain Inventory (BPI) | 6 months
  The BPI consists of questions related to pain intensity and pain interference on function. Responses for each item ranges from 0 (no pain) to 10 (pain as bad as you can imagine). Pain severity score (sum score of intensity items 1 to 4) and interference score (sum score of interference items 5 to 10) are reported. In addition, one item measure the localization of the most intense pain.
Semi-structured interview | 6 months
  The interview includes 32 items. Participants are asked about basic demographic information (e.g. years of education, occupation, living situation), medical conditions/ injuries (e.g. Have you ever been diagnosed with ADHD?), treatment/rehabilitation (e.g. Have you received cognitive rehabilitation?) and adverse life events (e.g. Have you lost a close family-member within the last 12 months?). In addition, participants are asked to describe challenges in their everyday life (e.g. Please tell me about challenges in your everyday life when it comes to achieving your goals, Do you easily get distracted from what you are doing?).

CONTACTS AND LOCATIONS:
Overall Officials: Magne Arve Flaten, phd prof, Study Director — Norwegian University of Science and Technology; Paul Georg Skogen, Study Director — St. Olavs Hospital, Clinic manager
Locations (3):
- Norway (3):
  - Oslo University Hospital - Rikshospitalet, Oslo
  - St. Olavs Hospital, Trondheim
  - Department of Psychology, Norwegian University of Science and Technology (NTNU), Trondheim

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Derived] Egset KS, Weider S, Hjemdal O, Ruud E, Hjort MA, Eilertsen MB, Sund AM, Stubberud J, Reinfjell T. Exploring the Discrepancy Between Subjective and Objective Measures of Executive Functions in Young Adult Survivors of Childhood Acute Lymphoblastic Leukemia. J Adolesc Young Adult Oncol. 2025 Aug;14(4):345-351. doi: 10.1089/jayao.2024.0105. Epub 2024 Nov 18. PMID 39552427